CLINICAL TRIAL: NCT02036931
Title: A Multicentre Observational Study to Evaluate Clinical Outcomes of the G7 Acetabular System
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: ORTHO.CR.GH20
Record Dates: First submitted 2014-01-14; First posted 2014-01-15 (Estimated); Results first posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Noninflammatory Degenerative Joint Disease; Rheumatoid Arthritis
Keywords: Joint; Osteoarthritis; Avascular Necrosis
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis; Osteonecrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Metal on Polyethylene articulation: G7 cup with Metal on Polyethylene articulation (MOP)
  Interventions: Device: Metal on Polyethylene articulation
- Ceramic on Polyethylene articulation: G7 cup with Ceramic on Polyethylene articulation (COP)
  Interventions: Device: Ceramic on Polyethylene articulation
- Ceramic on Ceramic articulation: G7 cup with Ceramic on Ceramic articulation (COC)
  Interventions: Device: Ceramic on Ceramic articulation

INTERVENTIONS:
Device: Metal on Polyethylene articulation — G7 Acetabular Cup System with Metal head on Polyethylene liner articulation (MOP)
  Other Names: MOP
  Groups: Metal on Polyethylene articulation
Device: Ceramic on Polyethylene articulation — G7 Acetabular Cup System with Ceramic head on Polyethylene liner articulation (COP)
  Other Names: COP
  Groups: Ceramic on Polyethylene articulation
Device: Ceramic on Ceramic articulation — G7 Acetabular Cup System with Ceramic head on Ceramic linear articulation (COC) - Outside the United States ONLY
  Other Names: COC
  Groups: Ceramic on Ceramic articulation

SUMMARY:
This is a prospective observational multi-center non-controlled study. The primary purpose of this study is to evaluate the clinical and radiographic performance of the G7 Acetabular Cup System.

DETAILED DESCRIPTION:
This is a prospective observational multi-center non-controlled study. The primary purpose of this study is to evaluate the clinical and radiographic performance of the G7 Acetabular Cup System in both primary and revision procedures, report safety and survivorship, and document instrument ease of use.

Preoperative and intraoperative data have been collected retrospectively and follow ups have been collected prospectively.

Clinical outcomes included the Harris Hip Score, Oxford Hip Score, and Radiographic Evaluations collected at 3 month, 1, 2 and 5 year follow-up time points. For the 7 and 10 year follow-up intervals, survivorship and adverse events have been collected.

ELIGIBILITY:
Inclusion Criteria:

* Noninflammatory degenerative joint disease including osteoarthritis and avascular necrosis
* Rheumatoid arthritis
* Correction of functional deformity
* Treatment of non-union, femoral neck fracture, and trochanteric fractures of the proximal femur with head involvement, unmanageable by other techniques
* Revision procedures where other treatment or devices have failed
* 18 years of age or older
* Subjects willing to return for follow-up evaluations

Exclusion Criteria:

* Infection, sepsis and osteomyelitis
* Subjects unable to cooperate with and complete the study
* Neurological conditions affecting movement
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2024-12 (Actual); Study Completion 2025-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Rohmer, Study Director — Zimmer Biomet
Locations (6):
- University Orthopedic Specialists, Tucson, Arizona, United States
- Clermont-Ferrand Hospital, Clermont-Ferrand, France
- University of Würzburg, Orthopedic, Würzburg, Germany
- Midwestern Regional Orthopaedic Hospital, Limerick, Ireland
- Reinier de Graaf Groep, Delft, Netherlands
- Hospital El Bierzo, Ponferrada, Spain

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metal on Polyethylene Articulation | Ceramic on Polyethylene Articulation | Ceramic on Ceramic Articulation
Started | 96 | 37 | 29
Completed | 37 | 15 | 10
Not Completed | 59 | 22 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metal on Polyethylene Articulation | Ceramic on Polyethylene Articulation | Ceramic on Ceramic Articulation | Total
Number analyzed (Participants) | 96 | 37 | 29 | 162
Age, Continuous [Mean (Full Range); unit: Years] | 68.8 [40 to 84] | 61 [40 to 83] | 61 [44 to 82] | 66 [40 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 26 | 7 | 79
  Male | 50 | 11 | 22 | 83
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Harris Hip Score [Mean (Standard Deviation); unit: Scores] — Population: Scores at preop visit are available for fewer patients than total enrollment due to retrospective data collection.
  Scores
    number analyzed (Participants) | 91 | 37 | 29 | 157
    (all) | 45.8 (16.7) | 43.1 (12.6) | 50.7 (15.4) | 46.1 (15.7)

OUTCOME MEASURES:

1. Primary Outcome: Harris Hip Score
Description: The Harris Hip Scale (HHS) is an outcome measure that includes a series of questions answered by the patient and physical examinations recorded by a qualified health care professional. The HHS covers four domains: pain (one item, 0-44 points), function and functional activities (seven items, 0-47 points), absence of deformity (one item, 0-4 points) and range of motion (one item, o-5 points). To obtain a final score, the points are summed. The outcome score can be categorized as Excellent:90 - 100; Good: 80 - 90; Fair: 70 - 80; Poor: < 70.
Time Frame: Pre-operative,1, 2, and 5 years postoperatively
Population: The number of participants decreased around the 5-year visit due to substantial patient loss at certain sites.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Metal on Polyethylene articulation | Ceramic on Polyethylene articulation | Ceramic on Ceramic articulation
Number analyzed (Participants) | 91 | 37 | 29
Score
  Pre-op | 45.8 (16.7) | 43.1 (12.6) | 50.7 (15.4)
  1 Year: number analyzed (Participants) | 76 | 30 | 26
  1 Year | 95.4 (7.4) | 94.2 (7.3) | 92.8 (10.0)
  2 Year: number analyzed (Participants) | 73 | 29 | 24
  2 Year | 96.1 (6.4) | 93.4 (9.5) | 94.3 (8.7)
  5 Year: number analyzed (Participants) | 31 | 13 | 21
  5 Year | 94.8 (7.1) | 91.7 (6.8) | 94.1 (7.8)

2. Secondary Outcome: Oxford Hip Score
Description: The Oxford Hip Score (OHS) is a patient-reported outcome measure that was developed to specifically assess the patient's perspective of outcome following THA. The OHS consists of twelve questions covering function and pain associated with the hip. To calculate the total score, each response is scored from 0 (worst outcome) to 4 (best outcome) and the sum of all 12 items is reported with a maximum of 48, representing the best score possible. The outcome score can be categorized as Excellent: > 41; Good: 34 - 41; Fair: 27 - 33; Poor: < 27.
Time Frame: Pre-op, 1, 2, and 5 years postoperatively
Population: The number of participants decreased around the 5-year visit due to substantial patient loss at certain sites.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Metal on Polyethylene articulation | Ceramic on Polyethylene articulation | Ceramic on Ceramic articulation
Number analyzed (Participants) | 87 | 37 | 26
Score
  Pre-op | 19.6 (9.1) | 16.2 (6.3) | 22.7 (9.0)
  1 Year: number analyzed (Participants) | 76 | 30 | 26
  1 Year | 46.1 (3.3) | 45.4 (3.3) | 45.4 (2.9)
  2 Year: number analyzed (Participants) | 73 | 29 | 26
  2 Year | 46.7 (2.4) | 45.2 (5.1) | 44.4 (6.1)
  5 Year: number analyzed (Participants) | 31 | 13 | 22
  5 Year | 46.5 (2.4) | 45.8 (2.4) | 43.4 (7.9)

3. Secondary Outcome: Survivorship
Description: Fraction of patients without a revision of any of the hip implant component, calculated with the Kaplan Meier (K-M) estimate.
Time Frame: 7 and 10 Year post-operative
Population: The K-M survival for CoP and CoC groups were only calculated up to 7 years because less than 20 cases remained at risk after that timepoint, which was below the level of detection to calculate a reliable Kaplan Meier estimate.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Metal on Polyethylene articulation | Ceramic on Polyethylene articulation | Ceramic on Ceramic articulation
Number analyzed (Participants) | 41 | 23 | 27
proportion of participants
  7 Year | 0.9762 [0.8428 to 0.9966] | 0.9697 [0.8037 to 0.9957] | 1.0000 [1.0000 to 1.0000]
  10 Year: number analyzed (Participants) | 39 | 16 | 13
  10 Year | 0.9762 [0.8428 to 0.9966] | NA — Below the level of detection (Only 16 cases remained at risk, which was insufficient [<20 cases] to calculate a Kaplan Meier estimate). | NA — Below the level of detection (Only 13 cases remained at risk, which was insufficient [<20 cases] to calculate a Kaplan Meier estimate).

4. Secondary Outcome: Survivorship
Description: as for outcome 3
Time Frame: 10 Year post-operative
Population: A Kaplan-Meier survival analysis was performed for all cases including 39 from MoP arm, 16 from CoP arm, 13 from CoC arm.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Entire Cohort: Entire Study Cohort
Arm/Group | Entire Cohort
Number analyzed (Participants) | 68
proportion of participants | 0.9818 [0.9277 to 0.9955]

5. Secondary Outcome: Radiographic Evaluation
Description: All radiographs have been reviewed by the investigators at each site in order to detect and report any abnormal and significant findings (including adverse events). The change from the angle of inclination between the different follow-ups is shown in the table.
Time Frame: Immediate post-op, 3 months, 1, 2, and 5 years
Population: The number of cases decreased around 5 years because two sites discontinued the study.
Measure: Mean (Standard Deviation); unit: Degree
Arm/Group | Metal on Polyethylene articulation | Ceramic on Polyethylene articulation | Ceramic on Ceramic articulation
Number analyzed (Participants) | 96 | 37 | 29
Degree
  Immediate Post-Op | 43.2 (5.8) | 41.9 (5.7) | 37.2 (6.1)
  3 Months: number analyzed (Participants) | 95 | 37 | 29
  3 Months | 42.8 (5.4) | 41.8 (5.5) | 37.2 (6.1)
  1 Year: number analyzed (Participants) | 77 | 30 | 26
  1 Year | 42.3 (5.7) | 42.4 (5.1) | 37.3 (6.3)
  2 Years: number analyzed (Participants) | 73 | 29 | 26
  2 Years | 42.7 (5.9) | 42.0 (5.4) | 37.6 (6.1)
  5 Years: number analyzed (Participants) | 31 | 13 | 19
  5 Years | 39.6 (4.3) | 41.8 (4.0) | 38.0 (6.9)

ADVERSE EVENTS:
Time Frame: Adverse events that met the criteria for serious adverse events (SAE), adverse device effects (ADE), serious adverse device effect (SADE), and unexpected serious adverse device effect (USADE) have been included throughout the participation of the study from date of surgery to 10-year follow-up.
Description: Adverse Events and Adverse Device Effects were documented during the whole course of the study.
Arm/Group | Metal on Polyethylene Articulation | Ceramic on Polyethylene Articulation | Ceramic on Ceramic Articulation
All-Cause Mortality (participants affected / at risk) | 5/96 | 1/37 | 3/29
Serious Adverse Events (participants affected / at risk) | 19/96 | 9/37 | 13/29
Other Adverse Events (participants affected / at risk) | 4/96 | 0/37 | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metal on Polyethylene Articulation (N=96) | Ceramic on Polyethylene Articulation (N=37) | Ceramic on Ceramic Articulation (N=29)
Revision (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) — ADE, Revision of Investigational Device
Dislocation (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 0 (0)
Death (unknown cause) (General disorders) | 5 (5) | 1 (1) | 3 (3) — Death from unknown cause - not reported in patient medical record
Infection (Infections and infestations) | 1 (1) | 2 (2) | 2 (2)
Liner wear (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal / Soft tissue (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
General AE (General disorders) | 9 (9) | 4 (5) | 6 (11)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metal on Polyethylene Articulation (N=96) | Ceramic on Polyethylene Articulation (N=37) | Ceramic on Ceramic Articulation (N=29)
Adverse Device Effects (ADE): Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2013-06-26): https://cdn.clinicaltrials.gov/large-docs/31/NCT02036931/Prot_000.pdf